CLINICAL TRIAL: NCT01964365
Title: An Open-label, Randomized, 6-Sequence, 3-Period Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between Rosuvastatin and Fenofibric Acid in Healthy Adult Subjects
Brief Title: Pharmacokinetics and Drug Interaction Study Between Rosuvastatin and Fenofibric Acid in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_DWJ1330001
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rosuvastatin (Experimental): multiple dose of Rosuvastatin 20mg
  Interventions: Drug: Cresto 20mg
- Fenofibric acid (Experimental): multiple dose of Fenofibric acid 135mg
  Interventions: Drug: Fenofibric acid 135mg
- Rosuvastatin + Fenofibric acid (Experimental): multiple dose of the combination of Rosuvastatin 20mg and Fenofibric acid 135mg
  Interventions: Drug: Cresto 20mg, Fenofibric acid 135mg

INTERVENTIONS:
Drug: Cresto 20mg — tablet, rosuvastatin 20mg
  Arms: Rosuvastatin
Drug: Fenofibric acid 135mg — capsule, fenofibric acid 135mg
  Arms: Fenofibric acid
Drug: Cresto 20mg, Fenofibric acid 135mg — rosuvastatin 20mg, Fenofibric acid 135mg
  Arms: Rosuvastatin + Fenofibric acid

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics profile and drug-drug interaction between rosuvastatin and fenofibric acid in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers aged 19 to 45 years
2. A sybject who has judged to be healthy by the investigator to participate in this study based on screening result
3. A subject who provided written informed consent to participate in this study and cooperative with regared to compliance with study related constraints

Exclusion Criteria:

1. A subject with sign or symptoms or previously diagnosed disease of liver, digestive system, cardiovascular, kidney, respiratory, endocrinology, neurology, immune system, hematology, and psychology function or other significant disease and history.
2. A subject who shows the following result in clinical laboratory test

   * AST, ALT > 1.25 times of the upper limit of normal range
   * PR ≥ 210 msec
   * QRS ≥ 120 msec
   * QT ≥ 500 msec
   * QTcF ≥ 500 msec
3. Subject who has taken other clinical medication from another clinical trial within 60-day period prior to the first administration of the study medication

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cmax | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
AUCtau | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods

SECONDARY OUTCOMES:
Cmin | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
Tmax | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
CL/F | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
T1/2 | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
Metabolic Ratio | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, Professor, Principal Investigator — BUSAN PAIK HOSPITAL
Locations (1):
- Inje University College of Medicine Busan Paik Hospital, Busan, South Korea